CLINICAL TRIAL: NCT00446316
Title: Effect of Antacids (Mg-Al-based) on Imatinib Mesylate (Gleevec®) Pharmacokinetics in Healthy Volunteers (CSTI571BUS257)
Brief Title: Effect of Antacids on Gleevec® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jan Beumer, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-088; CSTI571BUS257 (Other: Sponsor Protocol Number)
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Healthy volunteers; No condition; Pharmacokinetics study
MeSH Terms: interventions — Antacids; aluminum hydroxide, magnesium hydroxide, drug combination; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gleevec plus antacids (Experimental): Gleevec® will be administered at a dose of 400 mg, and the antacid (Maximum Strength Maalox®Max® Antacid/Anti-gas) at a dose level of 20 mL (equivalent to 1600 mg aluminum hydroxide and 1600 mg magnesium hydroxide). Half of the subjects will receive Gleevec® and antacid on day 15 and Gleevec® alone on day 1.
  Interventions: Drug: Antacids (Mg-Al-based); Drug: Imatimib Mesylate (Gleevec®)
- Imatimib Mesylate (Gleevec®) (Experimental): Gleevec® will be administered at a dose of 400 mg. Half of the subjects will receive Gleevec® and antacid on day 15 and Gleevec® alone on day 1. The other half will be treated in reverse order, i.e., they will receive the combination of Gleevec® and antacid on day 1, and Gleevec® alone on day 15. The antacids will be administered 15 minutes before the Gleevec® dose.
  Interventions: Drug: Imatimib Mesylate (Gleevec®)

INTERVENTIONS:
Drug: Antacids (Mg-Al-based) — the antacid (Maximum Strength Maalox®Max® Antacid/Anti-gas) at a dose level of 20 mL (equivalent to 1600 mg aluminum hydroxide and 1600 mg magnesium hydroxide).
  Other Names: Maalox
  Arms: Gleevec plus antacids
Drug: Imatimib Mesylate (Gleevec®) — Gleevec® will be administered at a dose of 400 mg. Half of the subjects will receive Gleevec® and antacid on day 15 and Gleevec® alone on day 1. The other half will be treated in reverse order, i.e., they will receive the combination of Gleevec® and antacid on day 1, and Gleevec® alone on day 15. The antacids will be administered 15 minutes before the Gleevec® dose.
  Other Names: Gleevec®

SUMMARY:
This is a research study that will investigate the effects of antacids (often used to treat stomach upset) on Gleevec® (a drug that is FDA-approved to treat some types of cancer) in healthy volunteers. Twelve healthy volunteers (six men and six women) will be recruited to complete the study. This research study will compare Gleevec® in the body when taken with and without antacids. Each volunteer will receive a 400 mg pill of Gleevec® on two occasions. One one occasion they will take the dose of Gleevec® alone. On another occasion, they will take the Gleevec® 15 minutes after taking a 20 mL dose of antacids. Several blood samples will be drawn to measure the concentrations of Gleevec® and its breakdown products in the blood, with and without the influence of antacids.

DETAILED DESCRIPTION:
This is an open-label, single-institution, randomized cross-over, fixed schedule study of the effects of Mg-Al-based antacids on Imatinib Mesylate (Gleevec®) pharmacokinetics. Healthy volunteers will be recruited to participate in this study such that twelve subjects (6 men / 6 women) will complete the study. Gleevec® pharmacokinetics will be assessed after oral administration of Gleevec® and after oral administration of Gleevec® with concomitant administration of magnesium-aluminum hydroxide-based antacid (Maalox). Gleevec® will be administered at a dose of 400 mg, and the antacid (Maximum Strength Maalox®Max® Antacid/Anti-gas) at a dose level of 20 mL (equivalent to 1600 mg aluminum hydroxide and 1600 mg magnesium hydroxide). Half of the subjects will receive Gleevec® and antacid on day 15 and Gleevec® alone on day 1. The other half will be treated in reverse order, i.e., they will receive the combination of Gleevec® and antacid on day 1, and Gleevec® alone on day 15. The antacids will be administered 15 minutes before the Gleevec® dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women 18 years of age or older. Healthy subjects are defined as individuals who are free from clinically significant illness or disease (such as coronary arterial disease, chronic heart failure, bleeding disorder, hypertension, chronic renal failure etc.) as determined by their medical history, physical examination, and laboratory studies.
* Body Mass Index (BMI) < 31 kg/m^2 (weight/height^2).
* Female subjects of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female subjects of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 7 days following discontinuation of study drug.
* Written, voluntary informed consent.
* Subjects participating in the protocol entitled "IRB: 0701014: Effect of Antacids (Mg-Al-based) on Imatinib Mesylate (Gleevec®) Pharmacokinetics in Healthy Volunteers (CSTI571BUS257) (UPCI #06-088)" will be eligible for participation in this study provided they meet all other eligibility criteria for this study.

Exclusion Criteria:

* Abnormal marrow function as defined by leucocyte, neutrophil, or platelet counts outside of normal limits.
* Any evidence of renal dysfunction (proteinuria; serum creatinine > upper limit of normal; or if serum creatinine > upper limit of normal, a calculated creatinine clearance < 60 mL/min/1.73 m2).
* Impaired hepatic function (liver enzymes greater than the upper limit of normal or bilirubin outside the normal range).
* Taking any medications (including over the counter products), herbal products, mineral supplements or vitamins (other than a daily multivitamin preparation), other than contraceptives (for women), within 2 weeks of start of the study. All forms of contraceptive medication are permissible for this study and would not result in a female's exclusion from participation. Patients who take medications on a chronic basis, such as antihypertensive medications or thyroid replacement therapy, etc. are not eligible for the study.
* Subjects that have received any other investigational agents within 28 days of first day of study drug dosing.
* Female subjects who are pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To define the effect of antacid administration on the pharmacokinetics (in particular the area under the Gleevec® plasma concentration versus time curve) of Gleevec® in healthy volunteers. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. Beumer, PharmD., PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute / Clinical and Translational Research Center (Hillman Cancer Center and Montefiore University Hospital locations), Pittsburgh, Pennsylvania, United States